CLINICAL TRIAL: NCT04489641
Title: Brief Group Psychotherapy for Anxiety and Depression: A Randomized Controlled Trial of Efficacy and Mechanisms of Change
Brief Title: Brief Group Psychotherapy for Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Jorge Corpas López, Clinical Professor, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Affective Disorder
MeSH Terms: conditions — Mood Disorders | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief group psychotherapy (Experimental): Group brief psychological intervention by adaptation of the Guide NICE "Common Mental Health Disorders" (ISBN 978-1-84936-585-7) and the unified protocol for the trasndiagnostic treatment of the emotional disorders of Barlow (Boisseau et al., 2010). This intervention is provided by clinical psychologist in primary care.
  Interventions: Behavioral: Psychological treatment
- Treatment as usual (TAU) (Active Comparator): Medication provided by a general practitioner.
  Interventions: Drug: Medication

INTERVENTIONS:
Behavioral: Psychological treatment — Psychological treatment
  Arms: Brief group psychotherapy
Drug: Medication — Pharmacological intervention
  Arms: Treatment as usual (TAU)

SUMMARY:
The present work aims to develop a randomized clinical trial with a sample of 100 patients diagnosed with anxiety and depression in primary care. All participants are tested by several self-reports related to emotional disorders in a repeated measures design, pre and post treatment. It is our aim this study will demonstrate that brief psychological treatments should be prioritized over pharmacological treatment in Primary Care. In addition, emotional regulation will be assessed and examined as a key factor in the clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety
* Depression

Exclusion Criteria:

* Severe mental disroders
* Drug abuse
* Suicidal ideation/severe depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety Disorder Assessment (GAD-7) | 12 weeks
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD.
The Patient Health Questionnaire (PHQ-9) | 12 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Beck Depression Inventory-Second Edition (BDI-II) | 12 weeks
  The BDI-II is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults. The BDI-II was revised in 1996 to be more consistent with DSM-IV criteria for depression. For example, individuals are asked to respond to each question based on a two-week time period rather than the one-week timeframe on the BDI. The BDI-II is widely used as an indicator of the severity of depression, but not as a diagnostic tool, and numerous studies provide evidence for its reliability and validity across different populations and cultural groups.
The Patient Health Questionnaire (PHQ-15) | 12 weeks
  It asseses somatoform symptoms. Scores could vary between 0-30 points.
Patient Health Questionnaire-Panic Disorder (PHQ-PD) | 12 weeks
  It measures panic disorder symotmos. Scores vould vary between 0-15 points.

SECONDARY OUTCOMES:
Emotional Regulation Questionnaire (ERQ) | 12 weeks
  It evaluates the tendency to regulate emotions. It consists of 10 items and participants have to respond according to a 7-points Likert scale. It has two subscales: reappraisal and suppression (six and four items respectively). The reappraisal subscale assesses the ability to change negative emotions while the suppression subscale assesses the tendency to repress and hide negative emotions.
Penn State Worry Questionnaire-Abbreviated (PSWQ-A) | 12 weeks
  It assesses the tendency to experience worry. It consists of eight items and patients have to respond according to a 5-point Likert-type scale.
Ruminative Response Scale-10 (RRS-10) | 12 weeks
  The RRS is the most used measure of rumination. The short version consists of 10 items that are responded on a 4-point Likert-type scale.
Metacognition Questionnaire-30 (MCQ-30) | 12 weeks
  This instrument has been used to assess metacognitive beliefs. It consists of 30 items that are responded on a 4-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Moriana, Principal Investigator — Universidad de Córdoba
Locations (1):
- Jorge Corpas, Córdoba, Andalusia, Spain